CLINICAL TRIAL: NCT05287360
Title: A Phase 1, Randomized, Open-label, Single-dose, Crossover Study to Evaluate the Bioequivalence of Four Formulations of Oral Rivoceranib Tablets in Healthy Subjects
Brief Title: A Study Comparing Four Different Rivoceranib Tablets in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elevar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RM-113
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Healthy
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence 1 (Experimental): Participants will receive rivoceranib on Day 1 of each period as a single dose under fasted conditions as follows:
  Period 1: Formulation 1; Period 2: Formulation 2; Period 3: Formulation 3; Period 4: Formulation 4
  There will be a washout period of 5 days between each dosing.
  Interventions: Drug: Rivoceranib
- Treatment Sequence 2 (Experimental): Participants will receive rivoceranib on Day 1 of each period as a single dose under fasted conditions as follows:
  Period 1: Formulation 2; Period 2: Formulation 4; Period 3: Formulation 1; Period 4: Formulation 3
  There will be a washout period of 5 days between each dosing.
  Interventions: Drug: Rivoceranib
- Treatment Sequence 3 (Experimental): Participants will receive rivoceranib on Day 1 of each period as a single dose under fasted conditions as follows:
  Period 1: Formulation 3; Period 2: Formulation 1; Period 3: Formulation 4; Period 4: Formulation 2
  There will be a washout period of 5 days between each dosing.
  Interventions: Drug: Rivoceranib
- Treatment Sequence 4 (Experimental): Participants will receive rivoceranib on Day 1 of each period as a single dose under fasted conditions as follows:
  Period 1: Formulation 4; Period 2: Formulation 3; Period 3: Formulation 2; Period 4: Formulation 1
  There will be a washout period of 5 days between each dosing.
  Interventions: Drug: Rivoceranib

INTERVENTIONS:
Drug: Rivoceranib — Rivoceranib will be supplied as film-coated tablets for oral administration as 4 different formulations: Formulation 1, 3, and 4 = 250 milligrams; Formulation 2 = 200 milligrams.
  Other Names: Rivoceranib Mesylate; Apatinib Mesylate

SUMMARY:
The main purpose of this trial is to compare a single dose of 4 different rivoceranib tablets in healthy adult participants.

DETAILED DESCRIPTION:
Participants will be randomized to 1 of 4 treatment sequences (1-4). Each participant will participate in 4 treatment periods. One formulation of rivoceranib will be administered per treatment period. Blood samples will be collected predose and up to 120 hours postdose to evaluate the pharmacokinetics (PK) of rivoceranib and its major metabolites.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a body mass index from 18.5 to 32.0 kilograms (kg)/meter squared (inclusive) and a weight of ≥ 50 kg at Screening.
2. Participants must be able to provide informed consent after risks and benefits have been explained. Participants must be capable of understanding, able to sign a written informed consent, and willing to comply with the protocol requirements.
3. Participants must agree to discontinue intake of beverages and foods known to interfere with cytochrome P450 (CYP) metabolic enzymes such as: grapefruit- and quinine-containing food and beverages (for example, tonic water, bitter lemon), orange juice, pomelos, cranberry, pomegranate, starfruit, Seville oranges (or marmalade made from them), garlic supplements or licorice, within 14 days prior to first dosing.
4. Participants must be in general good health as determined by the principal investigator (PI), based on pre-study medical and surgical history, physical examination, and clinical laboratory tests.
5. Participants must have normal blood pressure at Screening: systolic blood pressure < 130 millimeters of mercury (mmHg) and diastolic blood pressure < 85 mmHg.
6. Participants must have no clinically significant laboratory test results (≤ 1.5 x upper limit of normal for serum aspartate aminotransferase and alanine aminotransferase) at Screening.
7. Participants must have no clinically significant laboratory test results for prothrombin time, activated partial thromboplastin time, and international normalized ratio (> 20% outside the normal ranges) at Screening and Check-in.

Exclusion Criteria:

1. Participants who have participated in any investigational study within 30 days or 5 half-lives of the test drug's biologic activity, whichever is longer, prior to the first dosing.
2. Participants with any medical or surgical condition that may interfere with the absorption, distribution, or metabolism of the study drugs.
3. Participants who have a history of hypersensitivity to rivoceranib or any of its excipients.
4. Participants who are unwilling or unable to avoid xanthine- and caffeine-containing drinks (including many soft drinks, energy drinks, coffee, and tea) and foods (such as chocolate or coffee flavored) from 72 hours prior to first dosing.
5. Participants unable to refrain from or anticipate the use of:

   * any non-prescription medications, herbal remedies, or vitamin supplements within 14 days prior to the first dosing
   * any investigational drugs and prescription medications within 28 days prior to the first dosing. Use of any drugs or herbal remedies known to be significant inhibitors or inducers of CYP 3A4 and 2D6 enzymes for 28 days prior to the first dosing
   * appropriate sources (for example, Flockhart Table) will be consulted to confirm lack of PK/pharmacodynamic interaction with study drugs
6. Participants with corrected QT interval by Fridericia's formula > 460 microseconds or have clinically significant electrocardiogram findings, in the opinion of the PI, at Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Area Under The Concentration-time Curve From Time 0 To The Last Observed Non-zero Concentration (AUC0-t) For Plasma Rivoceranib And Its Major Metabolites | 0 (predose) up to 120 hours postdose
Area Under The Concentration-time Curve From Time 0 Extrapolated To Infinity (AUC0-inf) For Plasma Rivoceranib And Its Major Metabolites | 0 (predose) up to 120 hours postdose
Maximum Observed Concentration (Cmax) For Plasma Rivoceranib And Its Major Metabolites | 0 (predose) up to 120 hours postdose

SECONDARY OUTCOMES:
Percent Of AUC0-inf Extrapolated (AUC%extrap) For Plasma Rivoceranib And Its Major Metabolites | 0 (predose) up to 120 hours postdose
Apparent Volume Of Distribution During The Terminal Elimination Phase After Oral (Extravascular) Administration (Vz/F) For Plasma Rivoceranib | 0 (predose) up to 120 hours postdose
Apparent Total Plasma Clearance After Oral (Extravascular) Administration (CL/F) For Plasma Rivoceranib | 0 (predose) up to 120 hours postdose
Apparent First-order Terminal Elimination Half-life (t½) For Plasma Rivoceranib And Its Major Metabolites | 0 (predose) up to 120 hours postdose
Apparent First-order Terminal Elimination Rate Constant (Kel) For Plasma Rivoceranib And Its Major Metabolites | 0 (predose) up to 120 hours postdose
Time Of Observed Cmax (Tmax) For Plasma Rivoceranib And Its Major Metabolites | 0 (predose) up to 120 hours postdose
Participants Experiencing Treatment-emergent Adverse Events | Day 1 through Follow-up (14 days after the last dose of study drug)

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Tempe, Arizona, United States